CLINICAL TRIAL: NCT05241210
Title: Real-Time Feedback (RTFB) to Improve Colonoscopy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: we are on hold and may restart depending on a manual followed by automated assessment of existing files
Sponsor: University of Minnesota (Other)
Collaborators: University of Washington (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GI-2019-28090; DK106130 (Other Grant/Funding Number: University of Washington)
Record Dates: First submitted 2022-01-04; First posted 2022-02-15 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: Multiple successive arms testing new feedback options
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Testing of degree of mucosal inspection (Experimental): AI provides real-time feedback related to circumferential views during endoscope removal
  Interventions: Device: AI program for colonoscopy
- Testing of clearing of fecal debris (Experimental): AI provides real-time feedback related to removal of remaining fecal debris
  Interventions: Device: AI program for colonoscopy

INTERVENTIONS:
Device: AI program for colonoscopy — Provides real-time feedback on the endoscopist moniter during colonoscopy.

SUMMARY:
To test whether real-time feedback will improve quality of endoscopic examination.

ELIGIBILITY:
Inclusion Criteria:

- Any endoscopist willing to parcipate and performing routine colonscopy

Exclusion Criteria:

- No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4150 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adenoma Detection Rate | 5 months post procedure
  Percent change in ADR

CONTACTS AND LOCATIONS:
Overall Officials: Piet de Groen, MD, Principal Investigator — UMN
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No